CLINICAL TRIAL: NCT06152380
Title: Implementation of the Knee Care @Home Programme for Patients Recovering Anterior Cruciate Ligament Reconstruction: Protocol for a Randomised Feasibility Trial
Brief Title: Knee Care @Home Programme Feasibility Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Évora (Other)
Collaborators: Comprehensive Health Research Center (Other); Fundação para a Ciência e a Tecnologia (Other); Hospital da Misericórdia de Évora (Unknown)
Responsible Party: Principal Investigator, Joao Paulo Brites de Sousa, Auxiliar Professor, University of Évora
Other Study IDs: KC@H Feasibility
Record Dates: First submitted 2023-11-15; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Feasibility; Acceptability; Barriers; Facilitators; Anterior Cruciate Ligament Reconstruction; Internet-based Intervention; Exercise Therapy; Patient Satisfaction; Patient Engagement
MeSH Terms: conditions — Patient Satisfaction; Patient Participation | interventions — Exercise Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinic-based Rehabilitation: Individualised clinic-based face-to-face sessions with a physiotherapist in public or private rehabilitation facility
- Knee Care @Home: Individualised synchronous internet-based remote sessions at home via conferencing software under the supervision of a certified exercise and health coach as a complement to conventional clinic-based rehabilitation sessions.
  Interventions: Other: Knee Care @Home Programme

INTERVENTIONS:
Other: Knee Care @Home Programme — Over 24 weeks after undergoing surgical reconstruction of the anterior cruciate ligament, patients in the intervention group will receive supervised guidance on therapeutic exercises to be performed at home. This guidance will be provided through individualised synchronous internet-based remote sessions using conferencing software.
  Other Names: Synchronous internet-based remote sessions; Therapeutic Exercises
  Groups: Knee Care @Home

SUMMARY:
The main goal of this trial is to determine the feasibility of a randomized controlled trial for the Knee Care at Home Programme, rather than the effectiveness, for patients recovering from anterior cruciate ligament reconstruction. Specifically, the trial aims to: (1) assess the feasibility of studying the effectiveness of the Knee Care at Home programme, including patient engagement and satisfaction; and (2) conduct a qualitative assessment to identify barriers and facilitators in the implementation and delivery of the programme.

DETAILED DESCRIPTION:
Participants will be asked to take part in a 22-week intervention within a 24-week postoperative rehabilitation period following anterior cruciate ligament reconstruction. Internet-based remote sessions (3 times a week, 40 minutes per session) will supplement conventional clinic-based rehabilitation (face-to-face sessions). After the anterior cruciate ligament reconstruction, outcome measures are assessed during consultations with the orthopedic surgeon. These consultations occur after 4 weeks of intervention interval, except for the second postoperative consultation which occurs after a 2-week intervention period interval. Additional evaluations will occur during each remote session.

The team of researchers will evaluate the enrollment (screening, informed consent, eligibility, and allocation), data collection (response rates, missing data, and implementation and technical issues), intervention fidelity (adherence, adherence rate at remote sessions, adherence at conventional rehabilitation, quality of delivery, participant responsiveness, and safety), and acceptability (patient satisfaction and motivation).

ELIGIBILITY:
Inclusion Criteria

* Undergone primary ACLR regardless of surgical method and choice of autograft.
* Have a healthy contralateral (opposite) knee.
* The time between ACL injury and ACLR should not exceed 12 months.

Exclusion Criteria

* Declined to participate.
* Concomitant osteochondral injuries.
* Undergone multiple reconstructions of the lateral collateral ligament or posterior cruciate ligament.
* Significant lower limb injuries within the 12 months before the ACL injury.
* Medical conditions that may affect recovery.
* Using medication for mental disorders.
* Severe impairments in communication or balance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who have undergone anterior cruciate ligament reconstruction at Hospital da Misericórdia de Évora.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Enrolment: Screening | Preoperative consultation
  Quantitative data: The number of patients with anterior cruciate ligament injury who were approached and scheduled for anterior cruciate ligament reconstruction.
  Qualitative data: Open-ended questions posed to the orthopaedic surgeon regarding any ambiguities surrounding the screening procedure.
Enrolment: Informed Consent | Preoperative consultation
  Quantitative data: The number of patients who have signed the informed consent. Qualitative data: Open-ended questions posed to patients regarding their reasons for not signing the consent form.
Enrolment: Eligibility | First consultation after surgery (second week)
  Quantitative data: (1) The number of patients assessed for eligibility; (2) The number of patients meeting the inclusion criteria; and (3) The number of patients included.
  Qualitative data: (1) Open-ended questions to patients about the reasons for not participating; and (2) Open-ended question to orthopaedic surgeons about the reasons for patient ineligibility and enrollment ambiguities.
Enrolment: Allocation | First consultation after surgery (second week)
  Quantitative data: (1) The number of patients who agreed to be randomly assigned; and (2) The number of patients who dropped out after randomisation.
  Qualitative data: (1) Open-ended questions to patients about any problems they experienced with randomisation; and (2) Open-ended questions to orthopaedic surgeons about their reluctance to randomise patients.
Data Collection: Response rates | Up to 36 weeks postoperative
  Quantitative data includes the total number of outcome evaluation tools, the minutes spent using evaluation tools, and the number of unusable outcome measures.
Data Collection: Missing data | Up to 36 weeks postoperative
  Quantitative data includes the number of missing items.
Data Collection: Implementation and Technical issues | During each remote session, there will be a total of 22 weeks with 42 sessions between the 2nd and 24th postoperative week.
  Quantitative data: (1) Assessment of the costs and time allocated to resolving technical issues; and (2) Determination of the quantity of exercise and health coaches required to oversee patient recovery.
  Qualitative data: (1) Open-ended questions to patients regarding any technical issues encountered during remote sessions; and (2) Open-ended questions to exercise and health coaches regarding the adequacy of resources for remote sessions.
Intervention Fidelity: Adherence to the trial | During each orthopaedic consultation, there will be a total of 7 consultations on the 2nd, 4th, 8th, 12th, 16th, 20th, and 24th postoperative weeks, spanning a total of 22 weeks.
  Patients will be assessed in three areas: [1] withdrawal rate, including the number of patients who completed at least one remote session and then decided to withdraw, as well as the time point of withdrawal decision (quantitative data), and open-ended questions to those who withdraw to explain their reasons (qualitative data); [2] completion rate, which measures the number of patients that attend all remote sessions and consultations (quantitative data); and [3] follow-up rate, which measures the number of patients who remained in the study throughout the intervention period as a proportion of the total number of participants recruited at baseline (quantitative data).
Intervention Fidelity: Adherence rate at Remote sessions | During each remote session, there will be a total of 22 weeks with 42 sessions between the 2nd and 24th postoperative week.
  Areas: (1) General; (2) Consultations; (3) Compliance; and (4) Dosage.
  1. Open-ended questions will be asked to participants and coaches about reasons for absence from remote sessions (qualitative data).
  2. Data will be collected on completed evaluation consultations and duration (quantitative data). Open-ended questions will be asked to patients, surgeons, and assessors about reasons for non-compliance with evaluation consultations (qualitative data).
  3. Data will be collected on attendance, cancellations, lateness, logins, and completed remote sessions (quantitative data). Patient log sheets will be evaluated for qualitative data.
  4. Data will be collected on completed remote sessions, session parameters, exercises, and costs (quantitative data).
Intervention Fidelity: Adherence rate at Conventional Clinic-based Rehabilitation | During each orthopaedic consultation, there will be a total of 7 consultations on the 2nd, 4th, 8th, 12th, 16th, 20th, and 24th postoperative weeks, spanning a total of 22 weeks.
  Quantitative data: (1) Determine the number of patients participating in conventional clinic-based rehabilitation; (2) Track the number of sessions per week and their duration; and (3) Calculate the indirect costs associated with conducting the sessions.
  Qualitative Data: Open-ended questions posed to patients to gather information about the reasons for their absence from conventional clinic-based rehabilitation.
Intervention Fidelity: Quality of delivery | During each orthopaedic consultation, there will be a total of 7 consultations on the 2nd, 4th, 8th, 12th, 16th, 20th, and 24th postoperative weeks, spanning a total of 22 weeks.
  Quantitative data: Questions about the exercise and health coach's capacity to deliver the remote sessions.
  Qualitative data: Application of a questionnaire on an ordinal scale to patients about their self-rated level of agreement to statements about the exercise program using an 11-point Numeric Rating Scale (0 = strongly disagree and 10 = strongly agree).
Intervention Fidelity: Participant Responsiveness | During each remote session, there will be a total of 22 weeks with 42 sessions between the 2nd and 24th postoperative week.
  Quantitative data: (1) The number of exercises the patient was able to complete; and (2) The level of interest of patients in remote sessions based on previous criteria.
  Qualitative data: Application of a questionnaire on an ordinal scale to exercise and health coaches about their perception of the participant's effort during the remote sessions (SIRAS Scale).
Intervention Fidelity: Safety (adverse events) | During each remote session, there will be a total of 22 weeks with 42 sessions between the 2nd and 24th postoperative week.
  Quantitative data: (1) Assessing the frequency of signs and symptoms during remote sessions and between consultations; (2) Tracking the number of outcome measures showing no improvement or positive evolution; and (3) Recording the instances of exercise performance with excessive workload.
Acceptability: Satisfaction | During each orthopaedic consultation, there will be a total of 7 consultations on the 2nd, 4th, 8th, 12th, 16th, 20th, and 24th postoperative weeks, spanning a total of 22 weeks.
  Qualitative data: Patients will be asked to respond to some open-ended questions about their experience in remote sessions. These questions will be about: (1) attendance; (2) positive and negative consequences the intervention; and (3) other parameters about the intervention satisfaction it self. There will be a predetermined questionnaire on a Likert Scale, from 0=very dissatisfied, to 4=very satisfied regarding general satisfaction.
Acceptability: Motivation | During each orthopaedic consultation, there will be a total of 7 consultations on the 2nd, 4th, 8th, 12th, 16th, 20th, and 24th postoperative weeks, spanning a total of 22 weeks.
  Qualitative data: Participants are asked an open-ended question about their motivation to participate in the intervention using remote sessions.